CLINICAL TRIAL: NCT05164081
Title: DAICY Trial - Dual vs. Single-Antibiotic Impregnated Cement in Hemiarthroplasty for Femoral Neck Fracture: A Register-based Cluster-randomized Cross-over Controlled Trial
Brief Title: Dual vs. Single-Antibiotic Impregnated Cement in Hemiarthroplasty for Femoral Neck Fracture
Acronym: DAICY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DAICY
Record Dates: First submitted 2021-12-04; First posted 2021-12-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Femoral Neck Fractures; Prosthetic Infection
Keywords: femoral neck fracture; hip hemiarthroplasty; bone cement; antibiotic; periprosthetic joint infection; randomized controlled trial; dual impregnated antibiotic bone cement
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Gentamicins; gentamicin-polymethylmethacrylate bead; Cimetidine

STUDY DESIGN:
Intervention Model Description: Register-based cluster-randomized cross-over controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual antibiotic impregnated cement (Experimental): Patients treated with a cemented hip hemiarthroplasty using dual antibiotic loaded bone cement (gentamicin+clindamycin) COPAL G+C (Heraeus).
  Interventions: Combination Product: antibiotic loaded bone cement (gentamicin+clindamycin) COPAL G+C (Heraeus).
- Single antibiotic impregnated cement (Active Comparator): Patients treated with a cemented hip hemiarthroplasty using single antibiotic loaded bone cement (gentamicin) Paladins R+G (Heraeus) or Refobacin (Biomet).
  Interventions: Combination Product: antibiotic loaded bone cement (gentamicin) Paladins R+G (Heraeus) or Refobacin (Biomet).

INTERVENTIONS:
Combination Product: antibiotic loaded bone cement (gentamicin+clindamycin) COPAL G+C (Heraeus). — Hospitals are cluster-randomized to either arm for 2 years and then cross-over to the other arm for another 2 years.
  Arms: Dual antibiotic impregnated cement
Combination Product: antibiotic loaded bone cement (gentamicin) Paladins R+G (Heraeus) or Refobacin (Biomet). — antibiotic loaded bone cement (gentamicin) Paladins R+G (Heraeus) or Refobacin (Biomet).
  Arms: Single antibiotic impregnated cement

SUMMARY:
Rational for conducting the study: Periprosthetic joint infection (PJI) is the most feared complication following prosthetic replacement of the hip joint and is associated with increased mortality, morbidity and economic burden. The aim of the trial is to investigate whether the risk of periprosthetic joint infection after treatment with hemiarthroplasty performed due to femoral neck fracture is reduced after the use of dual-impregnated antibiotic loaded cement. The primary outcome variable is the incidence of periprosthetic joint infection within one year after the index procedure. Secondary outcome variables include the occurrence of re-operations for any reason, bacteriology, antibiotic treatment, mortality and health care costs.

DETAILED DESCRIPTION:
In Sweden, hip fractures annually affect close to 20,000 elderlies, often frail patients. Although the incidence of this injury seems to be stabilizing or even slightly declining, hip fractures cause an annual economic burden of no less than 800 million € in Sweden alone and the costs are increasing.

Femoral neck fractures (FNFs) are mainly a fragility fracture in the elderly and frail, predominantly affecting women after menopause but reports have indicated an increased incidence in elderly men. The average age of patients suffering a hip fracture has been increasing over the last decade and is around 80 years with an exponential increase of incidence with age. The lifetime risk of hip fracture in Sweden is 20% for women and 11% in men. A hip fracture is related to a doubled risk of death during the first year after fracture in comparison to age-matched controls.

FNFs are classified according to the degree of fracture displacement and the most widely used is the Garden classification. As displacement increases, the risk of disruption of the blood supply to the femoral head increases. Displaced fractures represent two thirds of the FNFs. With a disrupted vascular supply, the risk for healing disturbances, complications and reoperations increases when treated with internal fixation with screws or pins. For displaced fractures in elderly patients treated with internal fixation, failure rates of 35-50% have been reported in the literature. The most frequent complications are avascular necrosis and pseudarthrosis due to disrupted vascular supply of the femoral head and mechanical failure due to inadequate fixation. Long-term follow-up studies have emphasized the superiority of replacing the joint by hip arthroplasty in comparison to internal fixation in regard to hip function. Hip arthroplasty with either a total or hemiarthroplasty is a reliable option due to its ability to restore hip function and reduce the need for secondary surgery after an FNF. In hip arthroplasty implants are fixed to the bone with or without the use of bone cement (polymethyl methacrylate). Uncemented fixation in FNF patients has been linked to an increased risk for periprosthetic femoral fractures. In Sweden cemented hip arthroplasties are most frequently used and are regarded as the gold standard for FNF patients.

Bone cement or polymethyl methacrylate (PMMA) is widely used for implant fixation in orthopaedic procedures. PMMA acts as a void-filler that creates a tight space which holds the implant against the bone and acts as a 'grout'. Bone cements have no adhesive properties and rely instead on close mechanical interlock between the irregular bone surface and the prosthesis. PMMA is an acrylic polymer that is formed by mixing 2 sterile components, a liquid methyl methacrylate monomer and a powdered methyl methacrylate-styrene polymer. When mixed the liquid monomer polymerizes around the pre-polymerized powder particles to form hardened PMMA. An exothermic reaction generate heat in the process which reaches temperatures of around 82-86 °C in the body. In order to make the cement visible on radiographs, a contrast agent is added (zirconium dioxide or bariumsulphate).

Bone cement has proven useful as carrier of specific active substances, e.g., antibiotics added to the powder component. Antibiotics are delivered directly to the surgical site which in turn give a high concentration and low systemic concentration well below the clinical routine dosages for systemic single injections. Various antibiotics have been successfully mixed and used with bone cements like gentamycin, clindamycin etc. Compared to intramuscular administration, systemic concentration levels of gentamycin are low with bone cement, usual maximum concentrations below 1 μg/ml (<10%) without any detectable systemic levels after 7 days. In Sweden, antibiotic loaded cement is routinely used and represents the standard of care in cemented primary total hip arthroplasty, always in combination with systemic prophylaxis to reduce the risk for revision surgery due to periprosthetic joint infection (PJI). The type of antibiotic impregnated bone cement varies between regions, countries and type of surgical procedure performed.

In Sweden, the most commonly used cement is the low dose (≤ 2 g of antibiotic powder per 40 g cement) impregnated cement (Gentamycin). For revision procedures, a higher dose of gentamycin in combination with either vancomycin or clindamycin is often used and labelled dual-impregnated antibiotic cement (DIAC). For patients at risk for sustaining a PJI, i.e., hip fracture patients, some hospitals routinely use dual-impregnated antibiotic cement for hip arthroplasty procedures.

Surgical site infection (SSI) remains a severe complication linked to increased mortality, prolonged hospitalization, revision surgery, long-term treatment with antibiotics, dramatically increased costs and a strenuous rehabilitation. SSI is the third most commonly occurring healthcare-associated infection, accounting for 16% of reported infections. Rates of infection up to 7.3% for hemiarthroplasty have been reported. Parenteral antibiotics in elective primary total hip arthroplasty for osteoarthritis, have been shown to reduce SSI and antibiotic loaded cement, combined with systemic antibiotics is considered to be the most effective prophylaxis against infection. The potential of developing resistance among infecting organisms by using local antibiotics in general and especially DIAC has been under discussion but the clinical evidence remains sparse.

In a recent randomized study from England, the rate of infection following hemiarthroplasty for FNF was reduced from 3.5% with conventional single-impregnated antibiotic-loaded cement to 1.1% by using high-dose DIAC. Observational studies have indicated similar reduction in PJI. At present there is one ongoing large scale clinical (White 8) trial to further entangle the potential effect of DIAC in the United Kingdom.

Study design: Register-based, cluster randomized cross-over trial In the first step of the study, the orthopedic departments included are randomized to start with either the control or intervention treatment. After the first period of 2 years is completed, the study site will change to use the other treatment for the patients included in the following period of 2 years including a one month wash out period. At each department, information regarding the study is made available on the official web page, the orthopedic ward and the outpatient department.15 orthopedic department in Sweden has confirmed participation. All patients admitted and fulfilling the inclusion criteria and registered in the Swedish Fracture Registry or Swedish Arthroplasty Registry will be included. After the index surgery, procedural details and patient characteristics will be collected within the Swedish Arthroplasty Registry. Procedural details include type and brand of implant, type of components (uni- or bipolar head), type of cement (intervention: Dual-impregnated antibiotic bone cement or control: Single-impregnated antibiotic-laden bone cement), surgical approach and type of antibiotic prophylaxis. Patient characteristics registered in the Swedish Arthroplasty Registry include indication for surgery, age, sex, American Society of Anesthesiologists (ASA) grade and body mass index (BMI). Data on revision surgery performed and on reoperations are registered in the Swedish Arthroplasty Registry. Data on reoperations are also registered in the National Patient Registry. Mortality data are automatically available within the Swedish Fracture Registry and Swedish Arthroplasty Registry from the Swedish Drug Registry.

Study population: Patients aged ≥60 years

Number of patients: approx 7,000

Inclusion criteria:

* Age ≥60 years
* Diagnosis: Displaced femoral neck fracture type AO 31-B2 or B3/Garden type 3 or 4
* Eligible for hemiarthroplasty according to local guidelines and routines

Exclusion criteria:

* Previous inclusion of contralateral hip in the present study
* Pathological or stress fracture of the femoral neck, or fracture adjacent to a previous ipsilateral hip implant
* Unavailability of both interventions for a study participant (e.g., sensitivity to any of the components in the bone cement)
* Patients that have actively marked their hospital charts with an added privacy notice

Primary objective

1) The primary objective is to assess whether DIAC reduces the risk of PJI in patients with a femoral neck fracture treated with a HA by 50% within one year.

Secondary objective(s)

The secondary objective(s) of this study are to evaluate whether there is a difference between the intervention and control group in:

1. Any-reoperation at 1-year postoperatively.
2. Antibiotic prescription obtained from the Swedish Drug register at 120 days and 1-year post-surgery.
3. Mortality obtained from the Swedish Fracture Registry (SFR) within 90 days and 1-year post-surgery.

Other outcomes:

1. Resistance patterns of infections; all infections identified in the primary endpoint will be assessed for antibiotic resistance profiles. Identified in the NPR or SAR and obtained by assessing the medical files.
2. Resource use; cost data will be obtained from national databases or will be estimated in consultation with the hospital finance department at 120 days and 1-year post-surgery.

Trial period: Jan 1st 2022 - Jan 31st 2027

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Diagnosis: displaced femoral neck fracture type AO 31-B2 or B3/Garden type 3 or 4
* Eligible for HA according to local guidelines and routines

Exclusion Criteria:

* Previous inclusion of contralateral hip in the present study
* Pathological or stress fracture of the femoral neck, or fracture adjacent to a previous ipsilateral hip implant
* Unavailability of both interventions for a study participant (e.g., sensitivity to any of the components in the bone cement)
* Patients that have actively marked their hospital charts with an added privacy notice

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Periprosthetic joint infection | 1 year postoperatively
  The definition of PJI will be that the treating physicians defined presence of a PJI and started treatment (re-operation, or suppressive antibiotics, or combinations thereof).

SECONDARY OUTCOMES:
Any re-operation | 1 year postoperatively
  The rate of re-operation will be treated as a binary categorical variable, recorded together with an underlying time-to-event variable, and will be defined as the occurrence of any surgical procedure performed on the previously treated hip within one year after surgery.
Antibiotic suppression | 120 days and 1-year post-surgery
  Antibiotic prescription information will be obtained from the Swedish Drug Register.
Mortality | 90-day and 1-year mortality
  Occurrence of death (treated as a binary categorical variable), together with date and causes of death.

OTHER OUTCOMES:
The Resistance patterns of infections | 1 year postoperatively
  The rate of multiresistant bacterial strains in those patients with periprostetic joint infection; all infections identified in the primary endpoint will be assessed for antibiotic resistance profiles. The resistance profiles will be found at the microbiology department at the participating hospitals.
Cost-effectiveness | 1 year postoperatively
  Procedural costs for intervention and control treatment will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mukka, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sprowson AP, Jensen C, Chambers S, Parsons NR, Aradhyula NM, Carluke I, Inman D, Reed MR. The use of high-dose dual-impregnated antibiotic-laden cement with hemiarthroplasty for the treatment of a fracture of the hip: The Fractured Hip Infection trial. Bone Joint J. 2016 Nov;98-B(11):1534-1541. doi: 10.1302/0301-620X.98B11.34693. PMID 27803231
- [Background] Agni NR, Costa ML, Achten J, O'Connor H, Png ME, Peckham N, Dutton SJ, Wallis S, Milca S, Reed M. A randomized clinical trial of low dose single antibiotic-loaded cement versus high dose dual antibiotic-loaded cement in patients receiving a hip hemiarthroplasty after fracture: A protocol for the WHiTE 8 COPAL study. Bone Jt Open. 2021 Feb;2(2):72-78. doi: 10.1302/2633-1462.22.BJO-2020-0174. PMID 33630700
- [Background] Mukka S, Hailer NP, Moller M, Gordon M, Lazarinis S, Rogmark C, Ostlund O, Skoldenberg O, Wolf O; DAICY study group. Study protocol: The DAICY trial-dual versus single-antibiotic impregnated cement in primary hemiarthroplasty for femoral neck fracture-a register-based cluster-randomized crossover-controlled trial. Acta Orthop. 2022 Oct 5;93:794-800. doi: 10.2340/17453674.2022.4819. PMID 36200646
- See also: Study info site at the Swedish Fracture Registry home page — https://sfr.registercentrum.se/forskning/daicy/p/B1M6IVAFt